CLINICAL TRIAL: NCT07257263
Title: Exploring How Health Care Support Workers Respond to Distressed Behaviour in People With Dementia
Status: Active, not recruiting | Type: Observational
Sponsor: Royal Cornwall Hospitals Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2425.RCHT.44
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- staff

SUMMARY:
* To provide a narrative description of healthcare support workers experiences of responding to distressed behaviours in people with dementia
* To explore how these experiences might guide future training needs

ELIGIBILITY:
Inclusion Criteria:

* Healthcare support workers
* Working in a ward-setting caring for people with dementia
* Based in the main acute hospital

Exclusion Criteria:

* Registered staff (nurses and nursing associates)
* Allied Health Professionals and therapy support workers
* Healthcare support workers employed outside the main acute hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare support workers working in a ward-setting caring for people with dementia
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The study aims to capture the experiences of healthcare support workers caring for people with dementia that may display distressed behaviours | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Cornwall Hospitals Trust, Truro, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
To review with CI